CLINICAL TRIAL: NCT04188457
Title: Medical-economic Evaluation Comparing Intensive Outpatient Monitoring of Neuro-cardiovascular Diseases by Nurses, Doctors and Hospital and Private-sector Pharmacists, Compared to Usual Monitoring.
Acronym: DiVa
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: BEJOT Article 51
Record Dates: First submitted 2019-12-04; First posted 2019-12-06 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cerebrovascular Accidents; Myocardial Infarction
MeSH Terms: conditions — Stroke; Myocardial Infarction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Stroke - usual follow-up: Patient with either primary stroke, recurrent stroke, hemorrhagic, ischemic or Transient Ischemic Attack (TIA) with regular follow-up
  Interventions: Other: Usual follow-up
- Stroke - intensive follow-up: Patient with either primary stroke, recurrent stroke, hemorrhagic, ischemic or Transient Ischemic Attack (TIA) with intensive follow-up
  Interventions: Other: Intensive follow-up
- myocardial infarction - usual follow-up: Patient who has had a first or recurrent myocardial infarction with usual follow-up
  Interventions: Other: Usual follow-up
- myocardial infarction -intensive follow-up: Patient who has had a first or recurrent myocardial infarction with intensive follow-up
  Interventions: Other: Intensive follow-up

INTERVENTIONS:
Other: Usual follow-up — 2 medical consultations (nurse and doctor) over 24 months
  Groups: Stroke - usual follow-up; myocardial infarction - usual follow-up
Other: Intensive follow-up — 10 medical visits (nurse, doctor, pharmacist) over 24 months
  Groups: Stroke - intensive follow-up; myocardial infarction -intensive follow-up

SUMMARY:
Cerebral Vascular Accidents (stroke) and Myocardial Infarction (MI), which share the same risk factors, treatments and pathophysiological mechanisms, have become two major public health problems due to the increase in their prevalence rate and the longer survival after such an event in developed countries.

International data, including French data and data from our own registries, illustrate that:

* risk factors that are common, mainly hypertension, smoking, high cholesterol or diabetes, remain insufficiently controlled, although they are easily detectable and treatable;
* the incidence rate of stroke has doubled in 20 years in people under 55 years of age, increasing the number of people with chronic disabilities;
* 1-month and 1-year mortality rates for stroke and MIs have decreased by 17% in 5 years, increasing the number of survivors but with chronic disabilities;
* the aging of the population and the arrival of the baby boomers of the 1950s in the at-risk age groups has increased the at-risk population;
* Stroke and MI recurrence rates reached a threshold of 6% / year, in contrast to the very high rates of re-hospitalization at 1 year: 30% post-stroke and 20% post-MI, due to poorly anticipated and controlled complications. These reasons explain the lack of significant progress in preventing recurrences, preventable complications (heart failure and arrhythmias after MI; falls, sphincter and swallowing disorders, dementia and arrhythmias after stroke) and re-admission. This observation is aggravated by problems of medical demography and therefore the availability of neurologists, cardiologists and general practitioners.

Local and foreign experiments have demonstrated the value of intensive, coordinated and multi-professional stroke and MI monitoring, including nurses, in terms of: better control of risk factors and reduction of the rate of re-hospitalization by recurrence in stroke follow-up; improvement of the patient's general condition, control of risk factors, reduction in the number of events, decrease in the number of re-hospitalizations and their duration in MI follow-up. The value of pharmacists' additional intervention in intensive post-MI follow-up compared to routine follow-up has also been demonstrated, particularly in terms of significant improvement in patient compliance.

The hypothesis is that 2 years of intensive follow-up for both post-stroke or post-MI patients, by trained hospital and liberal nurses, in conjunction with doctors and pharmacists, is of medico-economic interest compared to usual follow-up. Therefore a medico-economic evaluation was designed to evaluate the efficiency of this model, which combines community-based and recourse care, prevention and coordination of care compared to usual follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient or legal representative who has given oral consent
* Patient over 18 years of age
* Patient with:

  * either a primary MI or a recurrent MI, not previously included, defined according to the criteria of the European Society of Cardiology and ICD-10
  * either a primary stroke, a recurrent stroke not previously included, hemorrhagic, ischemic or Transient Ischemic Attack (TIA), defined according to WHO criteria, the TOAST score and the ICD-10, with a Rankin score < 5.
* Patient followed up in one of the 6 public health establishments of the GHT 21-52 (regional group of hospitals) or at the Valmy clinic in Dijon also participating in the project
* Patient with estimated survival beyond 12 months

Exclusion Criteria:

* A patient who is not affiliated to the national health insurance system;
* A patient subject to legal protection (curatorship, guardianship)
* To be a patient subject to a measure of judicial safeguard;
* Pregnant, parturient or breastfeeding woman;
* Admitted for a condition other than stroke, TIA and MI;
* Experiencing heart failure before the MI;
* Be managed in EHPAD before and/or after stroke or IDM.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with stroke or myocardial infarction
Sampling Method: Non-Probability Sample
Enrollment: 859 (Actual)
Dates: Start 2020-10-15 (Actual); Primary Completion 2025-10-09 (Actual); Study Completion 2025-10-09 (Actual)

PRIMARY OUTCOMES:
Cost-utility ratio of the intensive monitoring strategy for each condition (stroke / myocardial infarction) | 24 month
  24-month incremental cost-utility ratio associated with the intensive post-stroke or post-MI follow-up strategy compared to the usual post-stroke or post-MI follow-up strategy, expressed as cost per year of life gained in good health (costs / QALY, score measured using EQ-5D-5L®).

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

IPD SHARING:
Plan to Share IPD: Yes
Relevant anonymized individual participant data that underlie the results reported in the articles resulting from this clinical trial will be shared to researchers who provide a methodologically sound proposal, to achieve aims of the approved proposal, upon reasonnable request to the principal investigator (Prof. Yannick Béjot, yannick.bejot@chu-dijon.fr). The data will become available after 3 months following the publication of the article and for 5 years.
Time Frame: The data will become available after 3 months following the publication of the article and for 5 years.
Access Criteria: request to the principal investigator (Prof. Yannick Béjot, yannick.bejot@chu-dijon.fr)

REFERENCES:
- [Derived] Bejot Y, Soilly AL, Bardou M, Duloquin G, Pommier T, Laurent G, Cottin Y, Vadot L, Adam H, Boulin M, Giroud M. Efficiency and effectiveness of intensive multidisciplinary follow-up of patients with stroke/TIA or myocardial infarction compared to usual monitoring: protocol of a pragmatic randomised clinical trial. DiVa (Dijon vascular) study. BMJ Open. 2023 Apr 26;13(4):e070197. doi: 10.1136/bmjopen-2022-070197. PMID 37185649